CLINICAL TRIAL: NCT00306085
Title: Autologous Bone Marrow Cell Treatment in Patients With Peripheral Atherosclerosis
Brief Title: Autologous Bone Marrow Cell Treatment in Peripheral Atherosclerosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Naples (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2006-03-14; First posted 2006-03-22 (Estimated); Last update posted 2006-03-22 (Estimated); Status verified 2006-03

CONDITIONS: Peripheral Vascular Diseases
Keywords: Peripheral arterial disease,; blood marrow cells,; therapeutic angiogenesis.
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease

INTERVENTIONS:
Genetic: Autologous bone marrow cells

SUMMARY:
Implantation of bone marrow cells, including endothelial progenitor cells, into ischemic limbs has been shown to improve collateral vessel formation. In the present study the safety and feasibility of autologous blood mononuclear cells implantation will be investigated in patients with severe peripheral atherosclerosis.Twenty cases will be enrolled. Improvement in the ankle-brachial pressure index (ABI:>0.1), ischemic ulcers and angiography as well as laser doppler flow will be evaluated until six months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of third or fourth class of peripheral atherosclerosis

Exclusion Criteria:

* Insuline dependent diabetes
* Cancer

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-04; Study Completion 2006-04

PRIMARY OUTCOMES:
Clinical and instrumental indexes of functional impairment of peripheral atherosclerosis.

SECONDARY OUTCOMES:
Angiographic and laser doppler measurements after six months from treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Sica, Study Director — University of Naples
Locations (1):
- University of Naples, Naples, Italy

REFERENCES:
- [Derived] Maione C, Botti C, Coppola CA, Silvestroni C, Lillo S, Schiavone V, Sica G, Sica V, Kumar V, Cobellis G. Effect of autologous transplantation of bone marrow cells concentrated with the MarrowXpress system in patients with critical limb ischemia. Transplant Proc. 2013 Jan-Feb;45(1):402-6. doi: 10.1016/j.transproceed.2012.10.031. PMID 23375329
- [Derived] Cobellis G, Botti C, Taddeo A, Silvestroni A, Lillo S, Da Ponte A, Villa ML, Sica V, Della Bella S. Successful bone marrow transplantation reveals the lack of endothelial progenitor cells mobilization in a patient with critical limb ischemia: a case report. Transplant Proc. 2010 Sep;42(7):2816-20. doi: 10.1016/j.transproceed.2010.04.047. PMID 20832596
- [Derived] Napoli C, Farzati B, Sica V, Iannuzzi E, Coppola G, Silvestroni A, Balestrieri ML, Florio A, Matarazzo A. Beneficial effects of autologous bone marrow cell infusion and antioxidants/L-arginine in patients with chronic critical limb ischemia. Eur J Cardiovasc Prev Rehabil. 2008 Dec;15(6):709-18. doi: 10.1097/HJR.0b013e3283193a0f. PMID 19050436